CLINICAL TRIAL: NCT00002092
Title: A Study to Evaluate the Effect of Cimetidine on CD4 Lymphocyte Counts in HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Community Research Initiative of New England (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 119A; 92-01
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Cimetidine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Cimetidine

INTERVENTIONS:
Drug: Cimetidine

SUMMARY:
To determine the change in CD4 count after 4 and 8 weeks in HIV-infected patients treated with cimetidine compared to placebo. To observe time-associated trends at weeks 4, 8, 12, and 16 in the change of CD4 counts for patients taking cimetidine for the full 16 weeks. To establish a safety record for cimetidine use in HIV-positive patients.

ELIGIBILITY:
Inclusion Criteria:

Concurrent Medication:

Allowed:

* All FDA-approved medications, antiretrovirals, and PCP prophylaxis drugs, with the exception of warfarin (Coumadin).
* Other self-prescribed medications available either over the counter or through buyer's clubs.

Patients must have:

HIV positivity.

NOTE:

* Patients on an antiviral or immunomodulating drug must have received it for at least 2 months and have no intention to make clinical or therapeutic changes in the first 8 weeks (such as adding a new agent or discontinuing effective viral suppressive therapy) that may interfere with the study.

NOTE:

* Patients who become pregnant after enrollment will be permitted to continue on study drug but must sign an additional informed consent indicating their awareness of the issues in taking a drug with limited safety data during pregnancy.

Prior Medication:

Allowed:

* Antiviral and immunomodulating drugs, provided patient has been on such therapy for at least 2 months prior to study entry.

Exclusion Criteria:

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known intolerance or hypersensitivity to cimetidine.
* Evidence of active opportunistic infection or malignancy requiring high-dose systemic chemotherapy.
* Any symptoms suggestive of concurrent illness that are not attributable to overall impairment by HIV or are not diagnosable based on the available evidence.
* Inability to swallow tablets (gastric feeding tubes are allowed).
* Not willing to comply with visit schedule and study procedures.

Concurrent Medication:

Excluded:

* Warfarin (Coumadin).

Prior Medication:

Excluded within 4 weeks prior to study entry:

* cimetidine (Tagamet), ranitidine (Zantac), famotidine (Pepcid), and nizatidine (Axid).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- CRI of New England, Brookline, Massachusetts, United States

REFERENCES:
- [Background] Cohen CJ, Hellinger JA, Day J, Salitsky N, Shevitz A, Zackin R, DeGruttola V. Lack of effect of cimetidine on lymphocyte subsets in patients infected with human immunodeficiency virus type 1. Clin Infect Dis. 1996 Nov;23(5):1049-54. doi: 10.1093/clinids/23.5.1049. PMID 8922801